CLINICAL TRIAL: NCT07152405
Title: A Phase III Randomized Controlled Clinical Study of BL-M07D1 for Injection Versus Investigator's Choice of Chemotherapy in Patients With HER2-positive Locally Advanced or Metastatic Gastric or Gastro-esophageal Junction (G/GEJ) Adenocarcinoma After Failure of First-line Anti-HER2 Therapy
Brief Title: A Study of BL-M07D1 Versus Investigator's Choice of Chemotherapy in Patients With HER2-positive Locally Advanced or Metastatic Gastric or Gastro-esophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-305
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-M07D1 (Experimental): Participants receive BL-M07D1 in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1
- Investigator's choice of chemotherapy (Active Comparator): Participants receive investigator's choice of chemotherapy in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Investigator's choice of chemotherapy

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: BL-M07D1
Drug: Investigator's choice of chemotherapy — Administration by intravenous infusion for a cycle of 2 or 3 or 4 weeks.
  Arms: Investigator's choice of chemotherapy

SUMMARY:
This trial is a registrational Phase III, randomized, controlled, open-label, multicenter study designed to evaluate the efficacy and safety of BL-M07D1 in patients with HER2-positive locally advanced or metastatic gastric or gastro-esophageal junction (G/GEJ) adenocarcinoma after failure of first-line anti-HER2 therapy and first-line standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. No gender restrictions;
3. Age at the time of signing the informed consent form is ≥18 years and ≤75 years;
4. Expected survival time ≥3 months;
5. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic HER2-positive gastric or gastroesophageal junction adenocarcinoma;
6. Must have at least one measurable target lesion as defined by RECIST v1.1;
7. ECOG performance status score of 0 or 1;
8. Toxicity from previous antitumor therapy has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
10. Organ function levels must meet the requirements;
11. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
12. Urine protein ≤2+ or <1000mg/24h;
13. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, and the serum pregnancy test must be negative. Patients must not be lactating. All enrolled patients (regardless of gender) should adopt adequate barrier contraception methods throughout the treatment cycle and for 7 months after the end of treatment.

Exclusion Criteria:

1. Received chemotherapy with mitomycin C and nitrosoureas within 6 weeks prior to the first dose, or underwent major surgery, radical radiotherapy, immunotherapy, etc., within 4 weeks prior to the first dose;
2. Previous treatment with HER2-ADC drugs, or ADC drugs with topoisomerase 1 inhibitors as the payload, or prior irinotecan therapy;
3. History of severe cardiovascular or cerebrovascular diseases within the past 6 months before screening;
4. Prolonged QT interval, complete left bundle branch block, third-degree atrioventricular block, or frequent and uncontrollable arrhythmias;
5. Concurrent pulmonary diseases resulting in severe impairment of lung function;
6. History of interstitial lung disease (ILD)/interstitial pneumonia requiring steroid treatment, or current ILD/interstitial pneumonia;
7. Diagnosis of other primary malignancies within 3 years prior to the first dose;
8. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg);
9. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (leptomeningeal metastases);
10. History of allergy to recombinant humanized antibodies or any excipient components of BL-M07D1;
11. History of autologous or allogeneic stem cell transplantation;
12. Unstable deep vein thrombosis requiring anticoagulant therapy during the screening period, or newly diagnosed deep vein thrombosis within 14 days;
13. Positive human immunodeficiency virus (HIV) antibody, active hepatitis B virus infection, or hepatitis C virus infection;
14. Occurrence of severe infections within 4 weeks prior to the first dose of the investigational drug; presence of infections requiring systemic treatment during the screening period;
15. Patients with massive serous cavity effusion, symptomatic serous cavity effusion, or poorly controlled serous cavity effusion;
16. Long-term systemic corticosteroid therapy (>10 mg/d prednisone or equivalent anti-inflammatory activity) or any form of immunosuppressive therapy within 2 weeks prior to randomization;
17. History of severe neurological or psychiatric disorders;
18. Presence of severe unhealed wounds, ulcers, or fractures within 4 weeks prior to signing the informed consent;
19. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks prior to signing the informed consent;
20. Conditions such as intestinal obstruction, Crohn's disease, ulcerative colitis, or chronic diarrhea;
21. Subjects planning to receive or having received live vaccines within 28 days prior to the first dose;
22. Presence of other severe physical or laboratory abnormalities, poor compliance, or any other factors that may increase the risk of participation in the study, interfere with study results, or make the patient unsuitable for participation in the study as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality